CLINICAL TRIAL: NCT07221916
Title: Stryker Customized Plates for Mandibular Reconstruction: A Retrospective Post Market Follow Up to Confirm Safety and Performance of Surgeon iD Mandible Reconstruction Plates
Brief Title: Stryker's Surgeon iD Mandible Reconstruction Plates: A Retrospective Post Market Follow Up
Acronym: SMRP
Status: Recruiting | Type: Observational
Sponsor: Stryker Craniomaxillofacial (Industry)
Responsible Party: Sponsor
Other Study IDs: Surgeon iD Plates _2023_01
Record Dates: First submitted 2025-07-31; First posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-08

CONDITIONS: Mandible Fracture; Mandibular Reconstruction
MeSH Terms: conditions — Mandibular Fractures | interventions — Mandibular Reconstruction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Mandibular Reconstruction — Mandibular Reconstruction or mandibular fracture fixation using a Surgeon iD Mandible Reconstruction Plate (referred to as Surgeon iD Plates).
  Other Names: Mandibular Fracture Fixation

SUMMARY:
A retrospective post market follow up to confirm safety and performance of Stryker's Surgeon iD Plates (SMRP) medical device. The study is performed to confirm the product's performance and safety by systematically collecting clinical data on its use.

DETAILED DESCRIPTION:
This is a retrospective non-interventional post-market follow up aiming at confirming safety and performance of Stryker's Surgeon iD Mandible Recon Plate when used in the clinical setting. This study will include patients who have previously undergone a surgical procedure involving the Study Device, with surgical outcomes evaluated retrospectively.

Based on a non-inferiority study power calculation a minimum of 27 patients will be enrolled in the study. Additional patients may be enrolled up to 80 subjects depending on site enrolment rate and patient availability. Up to 3 investigational sites within the United States and one in the EU will participate in this study. The primary outcome parameter evaluating successful reconstruction of the mandible without the need for unplanned revision surgery will be assessed at all available follow-up timepoints for included patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent primary or secondary mandibular reconstruction using a Stryker Surgeon iD Plate implant as per routine clinical practice.
2. Patients for whom data on the primary outcome variable is available.

Exclusion Criteria:

1. Patients with active local infections at the time of surgery.
2. Patients with known metal allergies and/or foreign body sensitivity at the time of surgery.
3. Potentially non-compliant patients who were unwilling or incapable of following post-operative care instructions.
4. Patients with inadequate bone quantity or quality necessary for plate fixation or stabilization at the time of surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients will be identified as having had a surgical procedure involving the Subject Device.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of successful reconstruction of the mandible without the need for unplanned revision surgery compared to benchmark devices in scientific literature. | Data collected at a single time point per patient in the course of 12 months
  Rate of unplanned revision surgery determined by reviewing adverse events in patient medical charts after surgery. Used to document whether an unplanned revision surgery was required or not for each patient.

SECONDARY OUTCOMES:
Infection rate | Data collected at time points from patient medical charts in the course of 12 months.
  Determined by adverse events reported from patient medical charts.
Intraoperative complications | Data collected at a single time point per patient in the course of 12 months.
  Determined by adverse events reported from patient medical charts.
Postoperative complications | Data collected at time points per patient in the course of 12 months.
  Determined by adverse events reported from patient medical charts.
Any known adverse events | Data collected at time points per patient in the course of 12 months.
  Determined by adverse events reported from patient medical charts.
Rate of Plate failure | Data collected at time points per patient in the course of 12 months.
  Determined by adverse events reported from patient medical charts.
Operating room (OR) time | Data collected at a single time point per patient in the course of 12 months.
  Time patients are operated (hh:mm)
Time to return to solid food/normal diet | Data collected at a single time point per patient in the course of 12 months.
  Time for patient to return to solid food/normal diet post operation (dd)
Rate of satisfactory occlusion achieved with orthodontic treatment. | Data collected at time points per patient in the course of 12 months.
  Assessed by review of individual patient medical records that document the rate of satisfactory occlusion achieved with orthodontic treatment.
Hospitalization time: ICU and normal ward | Data collected at a single time point per patient in the course of 12 months.
  Time the patient was hospitalized post procedure (dd:hh)
Short-form-12-health-survey-questionnaire (if available) | Data collected at time points per patient in the course of 12 months.
  Short-form-12-health-survey-Questionnaire (Scale of 0-100. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health).
Ischemia time | Data collected at a single time point per patient in the course of 12 months.
  Ischemia time (dd:hh)
EuroQol-5 Domain Questionnaire (if available) | Data collected at time points per patient in the course of 12 months.
  A descriptive system and a visual analogue scale (VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with three to five levels of severity. The VAS provides a subjective rating of overall health on a scale from 0 to 100 (higher is better)).
Facial Appearance, Quality of Life, and Satisfaction Questionnaire (if available) | Data collected at time points per patient in the course of 12 months.
  40 independently functioning scales and checklists. Multiple independent scales, each with a 0-100 score, where higher scores indicate better outcomes. Scores are calculated by summing responses on a 4-point Likert scale (e.g., strongly disagree to strongly agree), which are then converted to the 0-100 range. Each scale measures a specific aspect of facial appearance, quality of life, or adverse effects and cannot be summed into a single total score.

OTHER OUTCOMES:
Patient age | Data collected at a single time point per patient in the course of 12 months.
  Age (years)
Primary indication for the surgery / diagnosis | Data collected at a single time point per patient in the course of 12 months.
  Diagnosis collected from patient medical charts.
Follow-up time | Data collected at a single time point per patient in the course of 12 months.
  Post operative follow up time for patients within standard of care. Reported in patient medical charts during hospital follow up visit.
Surgical approach | Data collected at a single time point per patient in the course of 16 months.
  Surgical approach taken for the procedure. Including: transoral; transbuccal; submandibular; preauricular; other
Rate of osteotomy | Data collected at time points per patient in the course of 12 months.
  Cases where osteotomy (e.g. BSSO) was performed. Instrumentation used to perform the osteotomy.
Frequency of Maxilla-mandibular fixation | Data collected at time points per patient in the course of 12 months.
  Number of maxillo-mandibular fixation procedures (number per patient).
Relevant Medical conditions | Data collected at time points per patient in the course of 12 months.
  Descriptive data of any underlying medical conditions and medications recorded in patient medical charts that may be related to the device or primary outcome (qualitative measure).
Primary/secondary reconstruction performed | Data collected at time points point per patient in the course of 12 months
  Type of reconstruction procedure performed (e.g. immediately or after an initial surgery).
Localization of the defect | Data collected at time points point per patient in the course of 12 months.
  Area to treated by the device: mandibular ramus; mandibular body; mandibular condyle; parasymphysis; paramedian; other
Flap used | Data collected at a single time point per patient in the course of 12 months.
  Type of flap used: vascularized fibula flap, vascularized scapula flap, vascularized iliac crest flap, avascularized fibula flap, avascularized scapula flap, avascularized iliac crest flap, others
Radiation | Data collected at time points per patient in the course of 12 months.
  Exposure of patient to radiation therapy within 12 months around the surgery date recorded in patient medical charts. Radiation therapy performed on the anatomical area treated with the device. Any postoperative radiation therapy recorded in patient medical charts.
Dental reconstruction in a single stage surgery | Data collected at time points per patient in the course of 12 months.
  Data for dental reconstruction collected from patient medical charts.
Sterilization method used | Data collected at a single time point per patient in the course of 12 months.
  Sterilization method used for the device.
Fixation system used | Data collected at a single time point per patient in the course of 12 months.
  System used to fix the device during the procedure. Stryker Universal Mandible System; other Types and number of screws
Plate types | Data collected at a single time point per patient in the course of 12 months.
  2.0 or 2.8 plates used, hemi or full reconstruction plate used
Gender | Data collected at a single time point per patient in the course of 12 months
  Responses: Male, Female, undifferentiated, unknown
Patient height | Data collected at a single time point per patient in the course of 12 months.
  Height (cm, feet, inches)
Patient weight | Data collected at a single time point per patient in the course of 12 months.
  Weight (kg, lb)
Year smoking was stopped | Data collected at time points per patient in the course of 12 months.
  Year smoking was stopped (YYYY)
Smoking frequency | Data collected at time points per patient in the course of 12 month
  The frequency of exposure to smoking during periods of smoking (average number of cigarettes per day).
Smoking duration | Data collected at time points per patient in the course of 12 month
  Duration of smoking (pack years)
Years of active smoking | Data collected at time points per patient in the course of 12 month
  Total number of years active smoker (YY)

CONTACTS AND LOCATIONS:
Locations (2):
- UCSF Otolaryngology Head and Neck Surgery, San Francisco, California, United States
- Heinrich-Braun-Klinikum gGmbH, Zwickau, Germany

REFERENCES:
- See also: Kakarala, Kiran, Yelizaveta Shnayder, Terance T. Tsue, and Douglas A. Girod. 2018. "Mandibular Recon-struction." Oral Oncology. — https://pubmed.ncbi.nlm.nih.gov/29362116/
- See also: Lee,Z. et. al.2020. "The Latest Evolution in Virtual Surgical Planning: Customized Reconstruction Plates in Free Fibula Flap Mandibular Reconstruction." Plastic and Reconstructive Surgery. — https://pubmed.ncbi.nlm.nih.gov/32590512/
- See also: Witjes, Max J. H., Rutger H. Schepers, and Joep Kraeima. 2018. "Impact of 3D Virtual Planning on Recon-struction of Mandibular and Maxillary Surgical Defects in Head and Neck Oncology." Current Opinion in Otolaryngology and Head and Neck Surgery. — https://pubmed.ncbi.nlm.nih.gov/29470184/
- See also: Zeller AN, et al. Correction to: Patient-Specific Mandibular Reconstruction Plates Increase Accuracy and Long-Term Stability in Immediate Alloplastic Reconstruction of Segmental Mandibular Defects. J Maxillofac Oral Surg. 2022 Dec;21(4):1096. — https://pubmed.ncbi.nlm.nih.gov/36896089/
- See also: Möllmann HL, et al. Comparison of the Accuracy and Clinical Parameters of Patient-Specific and Conventionally Bended Plates for Mandibular Reconstruction. Front Oncol. 2021 Nov 26;11:719028. — https://pubmed.ncbi.nlm.nih.gov/34900674/
- See also: van Baar, et al, Accuracy of computer-assisted surgery in mandibular reconstruction: A systematic review. Oral Oncol. 2018 Sep;84:52-60. doi: 10.1016/j.oraloncology.2018.07.004. Epub 2018 Jul 20. PMID: 30115476. — https://pubmed.ncbi.nlm.nih.gov/30115476/